CLINICAL TRIAL: NCT06669039
Title: Comparison of Computer Controlled Intra-ligamentary Local Anesthesia and Conventional Inferior Alveolar Nerve Block in Primary Molars Extractions - Randomized Clinical Trail
Brief Title: Comparison of the Computer Controlled and Conventional Local Anesthesia Techniques in Primary Molar Extraction in Children Aged 5 to 9 Years Old
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Lamia Saleh AlGhamdi, Pediatric Dentist, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 109-05-23
Record Dates: First submitted 2024-10-28; First posted 2024-11-01 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Computer-controlled Intraligamentary Anaesthesia; Inferior Alveolar Nerve Block; Pain Perception; Anesthesia Effectiveness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional Inferior Alveolar nerve block (Active Comparator)
  Interventions: Procedure: Inferior Alveolar Nerve Block
- Computer-controlled Intraligamentary local anaesthesia (Experimental)
  Interventions: Device: Computer-controlled Local Anesthetic delivery system

INTERVENTIONS:
Device: Computer-controlled Local Anesthetic delivery system — Local anesthesia will be delivered using Computer-controlled Local Anesthetic delivery system.
  Arms: Computer-controlled Intraligamentary local anaesthesia
Procedure: Inferior Alveolar Nerve Block — Local anesthesia will be delivered using the conventional syringe
  Arms: Conventional Inferior Alveolar nerve block

SUMMARY:
The goal of this clinical trial is to assess pain perception, child stress level and compare the effectiveness between periodontal ligament anesthesia using Computer-controlled Local Anesthetic delivery system and the Conventional Inferior Alveolar Nerve Block during extraction of the primary molars.

The main questions it aims to answer are:

Is there a difference in pain perception, child stress level and anesthesia effectiveness between the CC-ILA system and the traditional syringe when administering IANB in pediatric patients undergoing primary molar extractions.

Researchers will compare CC-ILA system to traditional syringe when administering IANB to see if there a difference in pain perception, child stress level and anesthesia effectiveness.

Participants will:

Have their lower first primary molar extracted by receiving either periodontal ligament anesthesia using computer-controlled local anesthetic delivery system or the conventional inferior alveolar nerve bock.

Pain perception during the anesthesia process was measured using both objective criteria through the Sound-Eye-Motor scale and subjective assessment using Wong-Baker Faces Pain Rating Scale. Salivary cortisol level will be used to determine child stress level. The efficacy of anesthesia at various stages of the extraction procedure was evaluated using the Sound-Eye-Motor scale.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children (ASA I).
* Ranging in age from 5-9.
* Cooperative (Frankle ++).
* With mandibular first primary molars earmarked for removal owing to factors such as: extensive caries, crown damage, periapical lesions and unsuccessful pulp treatment.

Exclusion Criteria:

* Mobile teeth (Grade III).
* Ankylosed teeth.
* Teeth with root resorption (more than 1\3).
* Patients with facial cellulitis and when there is a need for supplemental anesthesia

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Pain | Immediately after receiving anesthesia
  Wong-Baker Faces Pain Rating Scale The scale contains a series of six faces ranging from a happy face at 0 to indicate "no hurt" to a crying face at 10 to indicate "hurts worst".
Pain | Immediately after receiving anesthesia
  Sound eye motor scale An observational scale uses child sound, eye and body movement to reflect on child comfort where score 1 reflect "comfort" and score 4 reflect "pain"
Stress level | Before and after local anesthesia delivery
  Child stress level after receiving either of anesthesia will be determined using salivary cortisol which will be collected by cortisol ELISA kit
Effectiveness | Through dental procedure
  Sound eye motor scale An observational scale uses child sound, eye and body movement to reflect on child comfort where score 1 reflect "comfort" and score 4 reflect "pain"

CONTACTS AND LOCATIONS:
Locations (1):
- King AbdulAziz University, Jeddah, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Pain perception scores, operator pain assessment scores and the anesthesia effectiveness scores.